CLINICAL TRIAL: NCT05871645
Title: Placenta Accreta Spectrum Management: Uterine Preservation Using JSICA Technique - Retrospective Cross-Sectional Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Amanda Rumondang, Principal Investigator, Dr Cipto Mangunkusumo General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-05-0541
Record Dates: First submitted 2023-02-27; First posted 2023-05-23 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Placenta Accreta
Keywords: JSICA technique; Placenta Accreta; Uterine Preservation
MeSH Terms: conditions — Placenta Accreta | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jakarta Surgical Uterine Conservation (JSICA) technique (Experimental): Cipto Mangunkusumo General Hospital's novel uterine preservation technique based on standard procedure
  Interventions: Procedure: Jakarta Surgical Uterine Conservation (JSICA) Technique
- Standard Hysterectomy (Active Comparator): Surgery to remove the uterus
  Interventions: Procedure: Standard Hysterectomy

INTERVENTIONS:
Procedure: Jakarta Surgical Uterine Conservation (JSICA) Technique — a. Identifying the placenta accrete site; b. Meticulous dissection to create a bladder flap; c. Incision 1 cm above the placenta accrete; d. Fetal delivery; e. Bottom incision to resect the placenta; f. Placental delivery; g. Uterus without placenta; h. The resection area is approximated using interrupted horizontal mattress suture; i. The continuous suture used to close all incision areas; j. Evaluation of uterine contraction
  Arms: Jakarta Surgical Uterine Conservation (JSICA) technique
Procedure: Standard Hysterectomy — The main types of hysterectomy are abdominal, vaginal, and laparoscopic hysterectomy
  Arms: Standard Hysterectomy

SUMMARY:
The goal of this study is to present the Jakarta Surgical Uterine Conservation (JSICA) technique and its perioperative outcomes in Placenta Accreta Spectrum patients. Participants are all patients undergoing standard hysterectomy or the Jakarta Surgical Uterine Conservation (JSICA) technique. Researchers will compare both groups to see if there are any differences in the perioperative outcomes.

DETAILED DESCRIPTION:
This study uses data from Cipto Mangunkusumo General Hospital's Placenta Accreta Case Register. This register includes all patients with a confirmed placenta accreta spectrum diagnosis. Data collected includes demographic characteristics, risk factors, surgery characteristics, and perioperative outcomes. In this study, researchers would like to evaluate the perioperative outcomes of the JSICA technique in comparison to a standard hysterectomy.

ELIGIBILITY:
Inclusion Criteria for JSICA:

1. Focal accreta invasion ( < 50% anterior wall)
2. Anterior invasion
3. No parametrial or bladder invasion
4. Residual tissue or healthy myometrium min 3 cm above the OUI or cervix
5. Good uterine contraction post-repair (with or without compression sutures)
6. Hemodynamically stable

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study apply for women with placenta accreta spectrum
Enrollment: 323 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Intraoperative bleeding | Perioperative
  Intraoperative bleeding in this study was measured by the amount of blood loss (cc) and classified into < 1.000 cc, 1.000-1.500 cc, and > 1.500 cc. .
Operation duration | Perioperative
  The operation duration was the time interval from skin incision to closure (hours) and classified into < 3 hours and > 3 hours.
Number of Patients Admitted to ICU | 24 hours
  ICU admission was identified by the documentation of number of patients' admission to the ICU
Rate of Intraoperative complications | Intraoperative
  Rate of intraoperative complications were identified by the documentation of injury to adjacent structures (bladder or ureter) or a need for transfusion.

SECONDARY OUTCOMES:
Intraoperative Bleeding in JSICA compared to hysterectomy | Perioperative
  Intraoperative bleeding in this study was measured by the amount of blood loss (cc) and classified into < 1.000 cc, 1.000-1.500 cc, and > 1.500 cc in comparison of JSICA to hysterectomy
Operation duration in JSICA compared to hysterectomy | Perioperative
  The operation duration was the time interval from skin incision to closure (hours) and classified into < 3 hours and > 3 hours in comparison of JSICA to hysterectomy
Number of Patients Admitted to ICU in JSICA compared to hysterectomy | 24 hours
  ICU admission was identified by the documentation of number of patients' admission to the ICU in comparison of JSICA to hysterectomy
Rate of Intraoperative complications in JSICA compared to hysterectomy | Perioperative
  Rate of intraoperative complications were identified by the documentation of injury to adjacent structures (bladder or ureter) or a need for transfusion in comparison of JSICA to hysterectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Maternal Fetal Medicine Division, Obstetric Gynecology Department Cipto Mangunkusumo General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No